CLINICAL TRIAL: NCT05842915
Title: Developing and Testing a Musculoskeletal National Audit in Community/Primary Care
Brief Title: The National Musculoskeletal Audit and Research Database
Status: Recruiting | Type: Observational
Sponsor: Keele University (Other)
Responsible Party: Sponsor
Other Study IDs: RG-0359-22
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Musculoskeletal Diseases
Keywords: Primary Care; Community; Benchmarking; Audit; Quality Improvement
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First Contact Practitioner (FCP): A continuous routine-data cohort study involving FCP primary care services aiming to recruit a minimum of 25patients per service from 10 FCP services, with complete data from at least 25 patients at baseline and 3-month follow up per service for each 12-month period. Data collection will involve:
  Patient survey (to collect outcomes and experiences)
  Organisational characteristics (collected via a survey to service leads and via publicly available national sources)
  Electronic health record (EHR) data (collected via a standardised FCP template and search within EHR systems)
  Interventions: Behavioral: Questionnaire
- MSK Community Services: A continuous routine-data cohort study involving MSK Community Services, aiming to recruit a minimum of 250 patients per service from a minimum of 10 MSK services, with complete data from at least 250 patients at baseline and 3-month follow up per service for each 12-month period. Data collection will involve:
  Patient survey (to collect outcomes and experiences)
  Organisational characteristics (collected via a survey to service leads and via publicly available national sources)
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Baseline and 3 month questionnaire

SUMMARY:
Developing and testing a musculoskeletal national audit in community/primary care

DETAILED DESCRIPTION:
This project aims to develop, setup and test an MSK national audit which will use patient and clinician inputted data to measure the quality of care for patients presenting in community MSK services and general practice with common MSK conditions. Secondly this project aims to use the national MSK audit information to understand and improve the quality and consistency of care for MSK patients.

ELIGIBILITY:
Inclusion Criteria:

(MSK Services)

* MSK service seeing adult (+18 years) set in community care
* MSK service with at least 10 WTE HCPs
* System in place for digital collection of PROM/PREM data

(FCP Services)

* FCP service seeing adult (+18 years) in primary care
* FCP service with at least 1 WTE FCP seeing MSK patients
* Use of EMIS or SYSTMONE
* Able to implement Midlands FCP template
* System in place for digital collection of PROM/PREM data

(For patients)

* +18 years
* Active phone number or verified email address to participate in the patient questionnaire
* Able to provide informed consent

Exclusion Criteria:

(MSK Services)

* Secondary care MSK services

(For patients)

* Has declined for data to be part of research as part of consent process
* Unable to complete surveys due to health issues including severe or terminal illness, severe learning difficulties or psychological disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 22,000 adult patients (over 2-year period), aged 18+ years consulting a) a Community MSK Service or b) a First Contact Practitioner (FCP) service in primary care, for a musculoskeletal pain condition
Sampling Method: Non-Probability Sample
Enrollment: 22000 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2028-06-07 (Estimated); Study Completion 2028-06-07 (Estimated)

PRIMARY OUTCOMES:
To provide a secure national MSK research database for participating MSK providers to upload their routinely collected data. | 12 months

SECONDARY OUTCOMES:
To develop a standard dashboard and reporting system that supports an ongoing automated process to analyse and present the data for quality improvement purposes. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Keele University, Keele, Staffordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No